CLINICAL TRIAL: NCT03052868
Title: Analysis of Neurocognitive Elements of Attention After Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SCCC-08111; STU 032011-207 (Other: UT Southwestern Medical Center)
Record Dates: First submitted 2017-02-09; First posted 2017-02-14 (Actual); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Cancer Nos
MeSH Terms: conditions — Neoplasms | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Data Collection (Other): The study visit will be scheduled for three to six months after completing adjuvant chemotherapy treatment. At the study visit, informed consent will be obtained and neurocognitive attention testing will be performed. The assessments chosen were carefully selected based on breadth, psychometric properties, standardized broad clinical use, good external validity and time efficiency. The testing time for the battery of neuropsychological tests is approximately 45-60 minutes. Participants will also be asked to complete a packet of several questionnaires including several self-rated measures of mood and quality of life, in addition to a brief questionnaire to obtain information about exercise, sleep, and education and employment backgrounds. It is estimated that questionnaire completion will require no more than 30 minutes. Participants will be seen on only one occasion, and may receive, upon request, written feedback about the results of the evaluation.
  Interventions: Other: Cognitive Assessment

INTERVENTIONS:
Other: Cognitive Assessment — Cognitive testing session

SUMMARY:
Data for this study will be obtained from the University of Texas Southwestern Medical Center Simmons Comprehensive Cancer Center. Participants will be recruited through Simmons Cancer Center. One hundred female breast cancer patients who have completed adjuvant chemotherapy will be enrolled. In order to reach this number, it is estimated that up to 125 eligible participants will need to be recruited. The study will last approximately two years. Participants will undergo one cognitive testing session, and each subject's total participation time will last no more than two hours.

DETAILED DESCRIPTION:
The study visit will be scheduled for three to six months after completing adjuvant chemotherapy treatment. At the study visit, informed consent will be obtained and neurocognitive attention testing will be performed. The assessments chosen were carefully selected based on breadth, psychometric properties, standardized broad clinical use, good external validity and time efficiency. The testing time for the battery of neuropsychological tests is approximately 45-60 minutes. Participants will also be asked to complete a packet of several questionnaires including several self-rated measures of mood and quality of life, in addition to a brief questionnaire to obtain information about exercise, sleep, and education and employment backgrounds. It is estimated that questionnaire completion will require no more than 30 minutes. Participants will be seen on only one occasion, and may receive, upon request, written feedback about the results of the evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Women;
* diagnosed with breast cancer Stages I-IV; and
* completed a treatment regimen of adjuvant chemotherapy three to six months prior to evaluation.

Patients may be receiving anti-hormonal treatment. All subjects will be native speakers of English who have a minimum of a high school education (or GED equivalent) in order to ensure the validity of the neuropsychological tests that will be administered. In order to limit age effects, participants will be between the ages of 40 and 70 years.

Exclusion Criteria:

* Subjects with a previous history of stroke, head injury with loss of consciousness greater than 30 minutes, major surgeries within the past 6 months unrelated to their breast cancer treatment, pre-cancer major Axis I psychiatric disorder, diagnosis of adult Attention Deficit Disorder, or other pre-existing disorder with known cognitive impairments (e.g. dementia, intellectual disability) will be excluded.
* Non- English speakers and subjects under the age of 40 or over the age of 70 will not be included.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Knowledge of cognitive outcomes of cancer treatment in breast cancer | 1 day
  battery of neuropsychological tests is approximately 45-60 minutes. Participants will also be asked to complete a packet of several questionnaires including several self-rated measures of mood and quality of life, in addition to a brief questionnaire to obtain information about exercise, sleep, and education and employment backgrounds

CONTACTS AND LOCATIONS:
Overall Officials: C. Munro Cullum, PhD, Principal Investigator — University of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: No